CLINICAL TRIAL: NCT04497077
Title: Comparison of Acute Tart Cherry Supplement Formulation and Dose on Inflammation and Oxidative Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Marywood University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 801765
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Inflammation; Oxidative Stress
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- single dose tart cherry capsule (Experimental): single dose tart cherry capsule
  Interventions: Dietary Supplement: tart cherry
- double dose tart cherry capsule (Experimental): double dose tart cherry capsule
  Interventions: Dietary Supplement: tart cherry
- single dose tart cherry juice (Experimental): single dose tart cherry juice
  Interventions: Dietary Supplement: tart cherry
- double dose tart cherry juice (Experimental): double dose tart cherry juice
  Interventions: Dietary Supplement: tart cherry
- single placebo capsule (Experimental): single placebo capsule
  Interventions: Dietary Supplement: placebo
- single placebo juice (Experimental): single placebo juice
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: tart cherry — Either tart cherry juice or freeze dried powdered tart cherry in capsule was given
  Arms: double dose tart cherry capsule; double dose tart cherry juice; single dose tart cherry capsule; single dose tart cherry juice
Dietary Supplement: placebo — either cornstarch capsule or kool-aid
  Arms: single placebo capsule; single placebo juice

SUMMARY:
A comparison of acute tart cherry formations (juice vs. powdered) and doses (single vs. twice daily) on inflammation and oxidative capacity.

DETAILED DESCRIPTION:
Participants will be randomly allocated to a group: one tart cherry capsule daily, two tart cherry capsules daily, one 8oz. bottle of tart cherry juice daily, two 8oz. bottles of tart cherry juice taken 8 hours apart, one placebo pill, and one 8oz. bottle of placebo. Participants will arrive to the lab at 8 am after an overnight fast of 10 hours. They will provide a blood sample and then ingest their study treatment. Participants will stay in the lab for a further 2 hours for additional blood draws then return to the lab in 6 hours for another blood draw. At this time if they are in a twice daily group they will receive their second treatment for the day. All participants will come back to the lab 24 hours later where they will give a blood sample and receive their next treatment. If they are in the twice daily group they will be provided with their next dose and given instructions to consume it in 8 hours. Participants will arrive 24 hours later for a final blood draw with no supplementation.

Blood samples will be measured pre-ingestion, 1 hour, 2 hours, 8 hours, 24 hours and 48 hours post-ingestion. Samples will be analyzed for plasma oxygen radical absorbance capacity (ORAC), uric acid (UA), and C-reactive protein (CRP).

ELIGIBILITY:
Inclusion Criteria:

* free of cardiovascular, metabolic and inflammatory conditions
* non-smokers
* no known allergy to cherries or cherry juice
* not be taking food supplements (turmeric/curcumin, cherry products, greens, etc.).

Exclusion Criteria:

* quit smoking less than one year ago.
* currently being treated for arthritis or an inflammatory condition.
* currently being treated for uncontrolled cardiovascular disease, high blood pressure, diabetes, fibromyalgia, or irritable bowel syndrome.
* pregnant.
* regularly consume cherries or are allergic to cherries or dairy.
* currently use anti-inflammatory medications,
* have used corticosteroids in the last two months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Change in c-reactive protein | 1 hour, 2 hours, 8 hours, 24 hours, and 48 hours post ingestion
  c-reactive protein (mg/L) measured via assay
Change in uric acid | 1 hour, 2 hours, 8 hours, 24 hours, and 48 hours post ingestion
  uric acid (mg/dL) measured via assay
Change in oxidative capacity | 1 hour, 2 hours, 8 hours, 24 hours, and 48 hours post ingestion
  oxygen radical absorbance capacity (uM Trolox equivalents) measured via assay

IPD SHARING:
Plan to Share IPD: No
upon request

REFERENCES:
- [Derived] Hillman AR, Uhranowsky K. Acute Ingestion of Montmorency Tart Cherry Reduces Serum Uric Acid but Has no Impact on High Sensitivity C-Reactive Protein or Oxidative Capacity. Plant Foods Hum Nutr. 2021 Mar;76(1):83-89. doi: 10.1007/s11130-021-00879-7. Epub 2021 Jan 27. PMID 33506357